CLINICAL TRIAL: NCT01539629
Title: Evaluation of Left Ventricular Autothreshold
Brief Title: ELEVATE (Evaluation of Left Ventricular Autothreshold) 3.0
Acronym: ELEVATE 3
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: ELEVATE 3.0
Record Dates: First submitted 2012-02-22; First posted 2012-02-27 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-10

CONDITIONS: Heart Failure
Keywords: Heart failure; Autothreshold; Pacing; CRT-D recipients; Left Ventricular evoked response signals
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pulse Width: One group reflecting two different pulse widths.
  Interventions: Device: Cardiac pacing

INTERVENTIONS:
Device: Cardiac pacing — Cadiac pacing via a pulse generator and implaned intracardiac leads.
  Other Names: COGNIS PG.

SUMMARY:
This 3rd phase of the ELEVATE study. The study is collecting data from an implanted CRT-D device to evaluate a new feature for future heart failure devices.

DETAILED DESCRIPTION:
ELEVATE 3.0 is an acute, prospective, multicenter feasibility study which is randomized within a patient test sequence and pulse width. The study is designed to characterize the performance of LVAT (Left Ventricular Authothreshold) feature.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are age 18 or above, or of legal age to give informed consent specific to state and national law
* Patients who have a COGNIS CRT-D device implanted for at least 24 hours, with or without an active right atrial lead
* Patients who have an active LV bipolar or unipolar lead
* Patients who have an active RV defibrillation lead
* Patients who are willing and capable of participating in all testing associated with this Clinical Investigation

Exclusion Criteria:

* Patients who have a COGNIS CRT-D that has less than or equal to one year of battery life remaining
* Patients who are pacemaker-dependent as defined as VVI 40 without intrinsic atrial or ventricular activity
* Patients who will not tolerate a pacing pause of up to 6 seconds
* Patients with a pre-existing unipolar pacemaker
* Patients who are unable or unwilling to maintain a supine or sitting position for 20-50 minutes
* Patients enrolled in any concurrent study, without Boston Scientific CRM written approval
* Women who are pregnant;women of childbearing potential must have a negative pregnancy test within 7 days prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be a sample of patients with COGNIS CRT-D devices.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-03; Primary Completion 2012-06 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Collect ventricular evoked response signal and CRT-D device data during LV only and Bi-Ventricular voltage step-down pacing. | Minimum of 24 hrs post CRT-D implant.
  The primary objective of this study is to collect real-time signals during LV pacing and voltage step-down from patients with implanted COGNIS devices.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth L Ellenbogen, MD, Principal Investigator — Virginia Commonwealth University Health System
Locations (4):
- United States (4):
  - Genesis Medical Center, Davenport, Iowa
  - Cardiology Consultants of Philadelphia, Yardley, Pennsylvania
  - Virginia Commonwealth University Health System, Richmond, Virginia
  - Wheaton Franciscan Health Care, Wauwatosa, Wisconsin